

Title: A Pivotal Phase 2 Trial of Ponatinib (AP24534) in Patients with Refractory Chronic Myeloid Leukemia and Ph+ Acute Lymphoblastic Leukemia

NCT Number: NCT01207440

SAP Approve Date: 14 December 2010

Certain information within this Statistical Analysis Plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable (PPD) information or company confidential information (CCI).

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

### STATISTICAL ANALYSIS PLAN

AP24534-10-201

PROTOCOL TITLE: A Pivotal Phase 2 Trial of Ponatinib (AP24534) in Patients with Refractory Chronic Myeloid Leukemia and Ph+ Acute Lymphoblastic Leukemia mia mia applicable applicable applicable

**PROTOCOL NUMBER:** AP24534-10-201

**IND NUMBER:** 78,375

**EudraCT NUMBER:** 2010-020414-28

ARIAD Pharmaceuticals, Inc **SPONSOR:** 

26 Landsdowne Street Cambridge, MA 02139-4234 Telephone: (617) 494-0400

Version 2.0 14 December 2010 **ORIGINAL ISSUE DATE:** 

### **REVISION/AMENDMENT HISTORY:**

| Amendme | nt Number | Version Number | Date |
|-------------------|-----------|----------------|------|
| | 60 | * | |
| | 7,0 | | |
| | ,01 | | |
| | 60 | | |
| Property of Takes | Ø. | | |
| 10 | > | | |
| 1 3/K | | | |
| 8 | | | |
| 0, | | | |
| 200 | | | |
| 0,0 | | | |

### TABLE OF CONTENTS

| 1 | Intr | oduction | ∠ |
|---|---|---|---|
| 2 | Stu | dy Objectives and Endpoints | 2 |
| | | udy Objectives | |
| | | Primary Objectives | |
| | | Secondary Objectives | |
| | 2.2 St | udy Design | Z |
| | 2.3 St | udy Endpoints | (O) |
| | 2 3 1 | Primary Endnoints | - 4 |
| | 2.3.2 | Secondary Endpoints | 5 |
| | 2.3.3 | Secondary Endpoints Exploratory Endpoints alysis Populations eated Population Cohorts A and D (CD CMI Potients) | <i>(</i> |
| 3 | Ana | alysis Populations | <i>6</i> |
| | 3.1 Tr | reated Population | <i>6</i> |
| | 3.1.1 | Cohorts A and B (CP CML Patients) | <i>6</i> |
| | 3.1.2 | Cohorts A and B (CP CML Patients) | <i>6</i> |
| | 3.2 Pe | er Protocol Population. | 7 |
| | 3.2.1 | Per Protocol (Cytogenetic) Population | 7 |
| | 3.2.2 | Per Protocol (Hematologic) Population | 7 |
| | 3.3 Sa | ifety Population | 7 |
| 4 | Sta | Per Protocol (Cytogenetic) Population Per Protocol (Hematologic) Population Ifety Population tistical Methods and Determination of Sample Size | 7 |
| | 4.1 De | etermination of Sample Size | 7 |
| | 4.1.1 | Cohorts A and B (Chronic Phase CML Patients) | 7 |
| | | Cohorts C-F (Accelerated Phase CML/Blast Phase CML/Ph+ ALL Patients) | |
| | 4.2 Sta | atistical Methods | 9 |
| | 4.2.1 | atistical MethodsDemographic and Baseline Characteristics | 9 |
| | 4.2.2 | Patient Disposition | 9 |
| | 4.2.3 | Patient Disposition Efficacy Analyses | 10 |
| | | .3.1 Primary Analysis of the Primary Endpoint | |
| | 4.2 | .3.2 Data Handling Rules for the Primary Analyses of the Primary Endpoint | |
| | 4.2 | .3.3 Sensitivity Analyses of the Primary Endpoint | |
| | 4.2.4 | Key Analyses of the Secondary Endpoints | 12 |
| | 4.2 | .4.1 Cohorts A and B (CP CML Patients) | 12 |
| | 4.2 | .4.2 Cohorts C-F (AP CML/BP CML/Ph+ ALL Patients) | |
| | 4.2 | .4.3 All Cohorts | 13 |
| | 4.2 | .4.4 Data Handling Rules for Secondary Endpoint Analyses | 13 |
| | | immaries of Data Handling Rules for Primary and Secondary Efficacy Analyses | |
| | | Subgroup Analyses of the Primary Endpoints and Key Secondary Endpoints | |
| | 4.3.2 | Treated Patients Not Eligible for Cohorts A-F | |
| | 4.3.3 | Safety Analyses | |
| $\bigcup_{X}$ | 4.3.4 | Study Drug Exposure | |
| | 4.3.5 | Exploratory Analyses | |
| 5 | Ref | ferences | 24 |

### LIST OF TABLES

| Table 1: | Planned Number of Patients for Each Cohort | |
|---|---|---|
| Table 2: | Sample Size Considerations for Each Cohort | |
| Table 3: | Patient Disposition | |
| Table 4:<br>Table 5: | Determination of PCyR With Assessment of < 20 Metaphases | |
| Table 6: | Summary of Data Handling Rules for Major Cytogenetic Response (MCyR) | 1 |
| | Summary of Data Handling Rules for Major Hematologic Response (MaHR) | 17 |
| Table 8: | Summary of Data Handling Rules for Analysis of Duration of Response† | |
| Table 9: | Summary of Data Handling Rules for Analysis of Major Molecular Response | 20 |
| | (MMR) | 21 |
| | Summary of Data Handling Rules for Major Hematologic Response (MaHR). Summary of Data Handling Rules for Analysis of Duration of Response (Summary of Data Handling Rules for Analysis of Major Molecular Response (MMR). | |
| | i kori | |
| Property of Taked | | |
| V1.0 14 Dece | ember 2010 | Page 3 |

#### 1 INTRODUCTION

Inis document specifies the statistical approaches and data handling conventions for key analyses that include the primary analyses for the primary endpoints and the analyses for key secondary endpoints.

2 STUDY OBJECTIVES AND ENDPOINTS

2.1 Study OF The Primary and Study OF The Primary endpoints and the analyses for key secondary endpoints. le applicable

#### 2.1 **Study Objectives**

#### 2.1.1 **Primary Objectives**

The primary objective of this trial is to determine the efficacy of ponatinib in patients with Chronic Myeloid Leukemia (CML) in chronic (CP), accelerated (AP) or blast phase (BP) or with Ph+ Acute Lymphoblastic Leukemia (ALL) who either are resistant or intolerant to either dasatinib or nilotinib or have the T315I mutation.

#### 2.1.2 **Secondary Objectives**

Secondary objectives are:

- 1. To further characterize the anti-leukemia activity of ponatinib in these patients as evidenced by clinical responses, molecular responses, and clinical outcomes
- 2. To characterize the molecular genetic status of patients
- 3. To examine the safety of ponatinib in these patients

#### **Study Design** 2.2

This is a phase 2, single-arm trial in patients with CML and Ph+ ALL. Table 1 summarizes the number of patients planned to be recruited in each cohort:

Table 1: Planned Number of Patients for Each Cohort

| ¢0 <sup>t</sup> | Chronic Phase (CP) | Accelerated<br>Phase (AP) | Blast Phase (BP)/Ph+ ALL | Total |
|---|---|---|---|---|
| Resistant/intolerant to | 100 | 40 | 40 | 180 |
| dasatinib or nilotinib | (Cohort A) | (Cohort C) | (Cohort E) | 180 |
| T315I mutation | 60 | 40 | 40 | 140 |
| (7.0 | (Cohort B) | (Cohort D) | (Cohort F) | 140 |
| Total | 160 | 80 | 80 | 320 |

Cohort A will consist of CP CML patients resistant or intolerant to dastinib or nilotinib. Cohort B will consist of CP CML patients with the T315I mutation. Cohorts C and E will consist of AP and BP/Ph+ ALL, respectively, who are resistant or intolerant to dasatinib or nilotinib. Cohorts D and F will consist of AP and BP/Ph+ ALL patients, respectively, with the T315I mutation.

Each of the 6 cohorts proposed in this trial are representative of distinct patient cohorts with licable Terms of Use different primary endpoints. Each cohort of patients will be analyzed separately for efficacy. The safety data from all cohorts will be pooled for the purpose of describing the safety of all treated patients as a whole. These cohorts can be viewed as 6 separate studies that are enrolled through a single "umbrella" protocol; therefore, no adjustments for multiplicity are planned.

#### 2.3 **Study Endpoints**

#### 2.3.1 **Primary Endpoints**

The primary endpoints for the cohorts are:

### **Cohorts A and B (CP CML Patients)**

Major cytogenetic response (MCyR), defined as complete cytogenetic response (CCyR) or Partial Cytogenetic Response (PCyR). Patients entering the trial already in PCyR must achieve a CCvR in order to be considered as achieving a MCyR. The criteria for response are provided in Attachment A of the protocol.

### **Cohorts C-F (AP CML/BP CML/Ph+ ALL Patients)**

Major hematologic response (MaHR), defined as complete hematologic response (CHR) and no evidence of leukemia (NEL). MaHR will be confirmed by a peripheral blood complete blood count (CBC) and differential no earlier than 28 days after the initial assessment of MaHR. The criteria for response are provided in Attachment A of the protocol.

#### **Secondary Endpoints** 2.3.2

Secondary endpoints for this trial are:

- Cohorts A and B: CHR as defined in Attachment A of the protocol.
- Cohorts C-F: MCyR.
- Confirmed MCyR, defined as 2 assessments of CCyR or PCyR at least 28 days apart. For CP patients entering the trial in PCvR, confirmed MCvR will be defined as 2 assessments of CCyR at least 28 days apart.
- Major Molecular Response (MMR) (as defined in Attachment A of the protocol).
- Duration of Response, defined as the interval between the first assessment at which the criteria for response were met until the criteria for progression (as defined in Attachment A of the protocol) are met, censored at the last date at which the criteria for response are met. An additional analysis will be performed in which patients who do not progress will be censored at the last dose of study drug. Duration of response will also be defined and analyzed as the time from the first assessment at which the criteria for response are met until the last assessment at which the criteria for response are met.
- Progression free survival, defined as the interval from the first dose of study treatment until the criteria for progression are met (as defined in Attachment A of the protocol) or death, censored at the last response assessment.
- Overall survival, defined as the interval from the first dose of study treatment until death, censored at the last date at which patient was known to be alive.

Time to response, defined as the interval from the first dose of study treatment until the criteria for response are first met, censored at the last assessment of response.

#### 2.3.3 **Exploratory Endpoints**

Exploratory endpoints for this trial are:



#### 3 ANALYSIS POPULATIONS

Each of the 6 cohorts will be analyzed separately. As stated in the protocol, patients will undergo testing at baseline for the presence of the T315I mutation via direct sequencing. The results of this test will determine the cohort to which a patient will ultimately be assigned.

For the purpose of statistical analyses, the following patient populations are defined for Cohorts A - F:

### 3.1

### 3.1.1

Cohorts A and B (CP CML Patients)

lation includes all patients assigning. Chronic phospad religions and religions are religious. This population includes all patients assigned to Cohort A or B who have received at least 1 dose of study drug. Chronic phase patients for whom a negative baseline T315I mutation result is received and who are resistant or intolerant to either dasatinib or nilotinib will be assigned to Cohort A. Chronic phase patients for whom a positive baseline T315I mutation result is received will be assigned to Cohort B. Patients who are not confirmed to have a detectable T315I mutation by direct sequencing but who are not resistant or intolerant to dasatinib or nilotinib (ie. who have been treated with only imatinib) will not be included in the treated population (or the per protocol population described below) and will be analyzed separately. We estimate that approximately 20% of patients with a history of a T315I mutation will have been treated with only imatinib, and thus will not be resistant or intolerant to dasatinib or nilotinib, and about onethird of these patients will lack the mutation by direct sequencing. We also estimate that this situation will most likely apply to the CP candidates, as patients with AP, BP and Ph+ALL will most likely have received more extensive therapy. Thus, we estimate that approximately 10 patients will fall into this group.

#### 3.1.2 Cohorts C-F (AP CML/BP CML/Ph+ ALL Patients)

This population includes all patients assigned to 1 of Cohorts C-F who have received at least 1 dose of study drug. CML patients in AP for whom a negative baseline T315I mutation result is received and who are resistant or intolerant to either dasatinib or nilotinib will be assigned to Cohort C. CML patients in AP for whom a positive baseline T315I mutation result is received will be assigned to Cohort D. CML patients in BP and Ph+ ALL patients for whom a negative baseline T315I mutation result is received and who are resistant or intolerant to either dasatinib

or nilotinib will be assigned to Cohort E. CML patients in BP and Ph+ ALL patients for whom a positive baseline T315I mutation result is received will be assigned to Cohort F. Patients who Terms of Use are not confirmed to have a detectable T315I mutation by direct sequencing and who are not resistant or intolerant to dasatinib or nilotinib will not be included in the treated population and will be analyzed separately, in the same fashion as described for Cohorts A and B.

#### 3.2 **Per Protocol Population**

#### 3.2.1 Per Protocol (Cytogenetic) Population

This population includes all patients in the treated population who have a baseline cytogenetic assessment with at least 20 metaphases examined. For Cohorts A and B (CP CML Patients), the primary analysis will be performed using the per protocol (cytogenetic) population. For Cohorts C-F (AP CML/BP CML/Ph+ ALL Patients), the analysis of the secondary endpoint of MCyR will be performed using the per protocol (cytogenetic) population.

#### 3.2.2 Per Protocol (Hematologic) Population

This population includes all patients in the treated population in Cohorts C-F who have a baseline BM assessment for which the percentage of BM blasts can be determined. For Cohorts C-F (AP CML/BP CML/Ph+ ALL Patients), the primary analysis will be performed using the per protocol (hematologic) population.

#### 3.3 **Safety Population**

This population includes all patients who have received at least 1 dose of study drug.

#### STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE 4

#### **Determination of Sample Size** 4.1

#### **Cohorts A and B (Chronic Phase CML Patients)** 4.1.1

As specified in Section 2.3, the primary endpoint for this trial for patients with CP CML (Cohorts A and B) is MCyR. MCyR rate is defined as the proportion of patients who have achieved a CCvR or PCvR after the initiation of study treatment. Patients entering the trial already in PCyR must achieve a CCyR in order to be considered as achieving a MCyR. As described above, the determination of PCyR status at baseline for the primary analysis will be based on an assessment with an examination of at least 20 metaphases.

The primary analysis of the primary endpoint of MCyR will be performed using a 2-sided exact 95% confidence interval (CI) for MCyR rate among all patients in the per protocol population in each cohort.

Data on the use of second generation tyrosine kinase inhibitors (TKIs) in patients who have failed dasatinib and nilotinib are available in several small studies (Giles, 2007; Quintas-Cardama, 2007; Garg, 2009), and we have used these data to estimate response rates in these historical control populations. These 3 studies demonstrate an approximately 30% MCyR in these patients. However, these are highly selected patient populations; they do not include patients who have failed more than 2 agents, and responses are typically of short duration. Thus for the purposes of this trial, the null or uninteresting MCvR rate is set at 20% for Cohort A

(resistant and intolerant CP patients). Here, and with regard to the cohorts discussed below, we intend that the specified null or uninteresting response rate defines a result that would not be clinically useful for the patient populations for which it is applicable. The alternative MCyR rate is set at 35% for Cohort A. The clinical implication of the alternative rate, in contrast, is that it would compare favorably with the historical experience for the specified patient populations and thus would be clinically beneficial. The overall alpha level for each cohort will be set at 0.05. With a cohort size of 100 patients, a minimum of 29 responders (ie, those with a CCyR and a PCyR) would need to be observed in Cohort A in order to observe an exact 95% CI such that the lower bound exceeds 20% and the upper bound exceeds 35%. Therefore, 100 patients will provide at least 85% power to distinguish between a null response rate of 20% and an alternative response rate of 35% in Cohort A. The study will also provide at least 98% power to distinguish between 20% and 40%, in which case 29 responses will also be required, and at least 78% power to distinguish between 30% and 45%, in which case 40 responses would be required.

With a cohort size of 100 patients, the maximum width of the exact 95% CI will be approximately 20% when the MCyR rate is in the expected range of 20% to 35%.

For Cohort B (T315I CP CML patients), the null or uninteresting MCyR rate is set at 10% and the alternative MCyR rate is set at 35%. Data on the use of second generation drugs (Garg 2009; Muller, 2009) in these patients suggest that less than 10% of patients achieve MCyR. With a cohort size of 60 patients, a minimum of 14 responders would need to be observed in Cohort B in order to observe an exact 95% CI such that the lower bound exceeds 10% and the upper bound exceeds 35%. Therefore, 60 patients will provide approximately 98% power to distinguish between a null response rate of 10% and an alternative response rate of 35% in Cohort B.

With a cohort size of 60 patients, the maximum width of the exact 95% CI will be 25% when the MCyR rate is in the expected range of 10% to 35%.

## 4.1.2 Cohorts C-F (Accelerated Phase CML/Blast Phase CML/Ph+ ALL Patients)

The sample sizes for Cohorts C to F (AP, and BP/Ph+ ALL) are based on similar considerations for each cohort (Garg, 2009). The endpoint for these cohorts is the MaHR. MaHR rate is defined as the proportion of patients achieving a CHR or NEL response. The null or uninteresting MaHR rate is set at 10% and the alternative MaHR 30%. With a cohort size of 40 patients, a minimum of 9 responders would need to be observed in Cohorts C to F in order to observe an exact 95% CI such that the lower bound exceeds 10% and the upper bound exceeds 30%. Forty patients in each cohort will provide approximately 89% power to distinguish between the null response rate of 10% and an alternative response rate of 30% in these cohorts.

The sample size considerations for each cohort are summarized in Table 2:

| Table 2: San | mple Size C | Considerations 1 | for Each Cohort |
|--------------|-------------|------------------|-----------------|
|--------------|-------------|------------------|-----------------|

| COHORT | Disease Phase | Eligibility | Primary | Sample Size | Effect Size | Power |
|---|---|---|---|---|---|---|
| | | Criterion | Endpoint | | | |
| A | CP | R/I | MCyR | 100 | 35% vs. 20% | ≥85% |
| | | | | | 40% vs. 20% | ≥98% |
| | | | | | 45% vs. 30% | ≥78% |
| В | CP | T315I | MCyR | 60 | 35% vs 10% | 98% |
| | | | | | 25% vs. 10% | 85% |
| C | AP | R/I | MaHR | 40 | 30% vs. 10% | 90% |
| D | AP | T315I | MaHR | 40 | 30% vs. 10% | 90% |
| E | BP/Ph+ALL | R/I | MaHR | 40 | 30% vs. 10% | 90% |
| F | BP/Ph+ALL | T315I | MaHR | 40 | 30% vs. 10% | 90% |

CP = chronic phase, R/I = resistance and/or intolerant, MCyR = major cytogenetic response, AP = accelerated phase, MaHR = major hematologic response, BP = blast phase, Ph+ ALL, Philadelphia chromosome positive acute ci io ine lymphoblastic leukemia.

#### 4.2 Statistical Methods

#### 4.2.1 **Demographic and Baseline Characteristics**

Demographic and baseline characteristics will be summarized separately for each cohort and will include at a minimum: age, gender, race, weight, country/region, and disease characteristics (eg, time since diagnosis, mutation status).

#### 4.2.2 **Patient Disposition**

Patient disposition will be summarized separately for each cohort. Table 3 below describes the anticipated presentation of key patient disposition categories for each cohort:

**Patient Disposition** Table 3:

| , cio | Treated Patients (N=) |
|-------------------------------------|-----------------------|
| Patients still on therapy | |
| Patients discontinued from therapy: | |
| In survival follow-up | |
| Died | |
| Lost to follow-up | |
| Withdrew consent | |
| Primary reason for discontinuation | |
| Progressive Disease | |
| Adverse Event | |
| Death | |
| Consent withdrawn | |
| Noncompliance with study drug | |
| Protocol violation | |
| Physician decision | |
| Lack of Efficacy | |
| Lost to follow-up | |
| Pregnancy | |
| Withdrawal by subject | |
| Other | |

Soluse

### 4.2.3 Efficacy Analyses

### 4.2.3.1 Primary Analysis of the Primary Endpoint

### **Cohorts A and B (CP CML Patients)**

As specified in Section 2.3, the primary endpoint for patients with CP CML in Cohorts A and B is MCyR. MCyR rate is defined as the proportion of patients who have achieved a CCyR or PCyR after the initiation of study treatment. Patients entering the trial in PCyR must achieve a CCyR in order to be considered as achieving a MCyR. Specifically, Table 4 summarizes how patient MCyR status will be classified based on baseline cytogenetic assessment:

Table 4: MCyR Classification and Baseline Cytogenetic Assessment

| | On-Study Assessment | | |
|----------------------------|---------------------|------|----------------|
| <b>Baseline Assessment</b> | PCyR | CCyR | Less than PCyR |
| Less than PCyR | MCyR | MCyR | No MCyR |
| PCyR | No MCyR | MCyR | No MCyR |

PCyR = partial cytogenetic reponse, CCyR = complete cytogenetic response, MCyR = major cytogenetic response.

The primary analysis of the primary endpoint will be performed using an exact 95% CI for the MCyR rate, using the per protocol (cytogenetic) population for each cohort. Patients who do not meet the criteria for MCyR will be analyzed as non-successes.

### Cohorts C-F (AP CML/BP CML/Ph+ ALL Patients)

The primary endpoint for patients with AP or BP CML or patients with Ph+ ALL in Cohorts C – F is MaHR. MaHR rate is defined as the proportion of patients who have achieved a CHR or NEL response after the initiation of study treatment.

The primary analysis of the primary endpoint will be performed using an exact 95% CI for the MaHR rate using the per protocol (hematologic) population for each cohort. Patients who do not meet the criteria for MaHR will be analyzed as non-successes.

### **All Cohorts**

In the event of over-enrollments beyond 10% of the planned sample size, a sensitivity analysis will be performed on the per protocol population when the sample size requirement is first realized.

The 6 cohorts will be analyzed separately and no adjustments for multiplicity are planned.

## 4.2.3.2 Data Handling Rules for the Primary Analyses of the Primary Endpoint

The key data handling rules for the primary efficacy analyses are as follows:

- All CP CML patients (Cohorts A and B) will have an opportunity to demonstrate MCyR up to 12 months after initiation of study treatment. Patients in Cohorts A and B who do not respond by 12 months after the initiation of study treatment will be analyzed as non-successes.
- All AP/BP phase CML patients and Ph+ ALL patients (Cohorts C, D, E and F) will have an opportunity to demonstrate MaHR up to 6 months after initiation of study treatment. Patients

in Cohorts C-F who do not respond by 6 months after the initiation of study treatment will be analyzed as non-successes.

- For patients entering the trial in less than PCyR, determination of MCyR requires a cytogenetic assessment with at least 13 metaphases examined:
  - o If 20 or more metaphases are examined, determination of MCyR will be based on the %Ph+ cells as specified in Attachment A of the protocol.
  - If 13-19 metaphases are examined, determination of MCyR will be performed as follows:

**Table 5:** Determination of PCyR With Assessment of < 20 Metaphases

| Number of<br>metaphases<br>examined | ≤12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 |
|---|---|---|---|---|---|---|---|---|
| Number of Ph+<br>cells | Any<br>Number | 0 | ≤1 | ≤2 | ≤3 | <b>4</b> | ≤5 | ≤6 |
| % Ph+ | | 0% | ≤7% | ≤13% | ≤19% | ≤24% | ≤28% | ≤32% |
| Response | Not<br>Evaluable* | PCyR | PCyR | PCyR | PCyR | PCyR | PCyR | PCyR |

\*The minimum of 13 metaphases is based on the threshold for MCyR of 7 Ph+ cells out of 20 metaphases.

- For patients entering the trial in PCyR, a CCyR must be observed in order to meet the criteria for MCyR; therefore, determination of MCyR requires a cytogenetic assessment with at least 20 metaphases examined.
- The criteria for initial determination of MaHR require the following sources of data:
  - o BM Aspirate,
  - o CBC with Differential,
  - Physical Exam.

In order to meet the criteria for MaHR, the above assessments must be performed within 14 days of one another. At assessments subsequent to the assessment at which the criteria for MaHR are first met, a physical exam is not required.

- Initial determination of MaHR must be confirmed no earlier than 28 days later; this confirmation requires the following source of data:
  - o CBC with Differential.

# 4.2.3.3 Sensitivity Analyses of the Primary Endpoint

Two additional sensitivity analyses of the primary endpoint will be performed as follows:

### **Sensitivity Analysis 1**

Sensitivity Analysis 1 is intended to assess the impact of the use of the per protocol population and the timing of when patients first demonstrate the criteria for success.

- Analysis of the primary endpoint will be performed on the treated population as specified in Section 3.
- For analyses of MCyR (primary endpoint for Cohorts A and B), all patients in the treated population will be included, regardless of the number of metaphases examined for the baseline cytogenetic assessment.
- The determination of PCyR status at baseline will be based on the percentage of Ph+ cells, regardless of the number of metaphases examined.
- Determination of success/not a success will be based on all available data in the database, regardless of when the criteria for success are met.

### **Sensitivity Analysis 2**

Sensitivity Analysis 2 is intended to assess the impact of patients for whom the baseline T315I direct sequencing result is not received until after the first bone marrow assessment.

- Patients for whom a **positive** baseline T315I direct sequencing result is received after the first cytogenetic response assessment (CML patients in CP) or BM assessment (CML patients in AP or BP and Ph+ ALL patients) will be analyzed as T315I-.
- Patients for whom a **negative** baseline T315I direct sequencing result is received after first cytogenetic response assessment (CML patients in CP) or BM assessment (CML patients in AP or BP and Ph+ ALL patients) will be analyzed as T315I+.
- For analyses of MCyR (primary endpoint for Cohorts A and B), all patients in the treated population will be included, regardless of the number of metaphases examined for the baseline cytogenetic assessment.
- The determination of PCyR status at baseline will be based on the percentage of Ph+ cells, regardless of the number of metaphases examined.
- Determination of success/not a success will be based on all available data in the database, regardless of when the criteria for success are met.

### 4.2.4 Key Analyses of the Secondary Endpoints

The key analyses of the secondary endpoints are specified below. Data handling rules for these analyses are specified in Section 4.2.4.4

### 4.2.4.1 Cohorts A and B (CP CML Patients)

• CHR the CHR rate is defined as the proportion of patients who have achieved a CHR after the initiation of study treatment. Chronic phase CML patients entering the trial in CHR will be excluded from this analysis. The analysis will be performed using a 2-sided exact 95% CI for the CHR rate.

### 4.2.4.2 Cohorts C-F (AP CML/BP CML/Ph+ ALL Patients)

• MCyR: the MCyR rate is defined as the proportion of patients who have achieved a CCyR or PCyR after the initiation of study treatment. The analysis will be performed using a 2-sided exact 95% CI for the MCyR rate, using the per protocol population.

### **4.2.4.3 All Cohorts**

- Confirmed MCyR: the confirmed MCyR rate is defined as the proportion of patients who
  have achieved a confirmed CCyR or PCyR after the initiation of study treatment. Patients
  entering the trial already in PCyR must achieve a confirmed CCyR in order to be considered
  a success for the confirmed MCyR rate. The analysis will be performed using a 2-sided
  exact 95% CI for the confirmed MCyR rate.
- Duration of response will be estimated using the Kaplan-Meier method. The median duration of response and 95% CI will be calculated. An additional analysis will be performed defining the duration as the time from the first assessment at which the criteria for response are met until the last assessment at which the criteria for response are met. Duration of response will be analyzed for MCyR, MaHR (Cohorts C-F), CHR (Cohorts A and B), and MMR.
- Progression-free survival, overall survival and time to response will be estimated using the Kaplan-Meier method. The median progression-free survival, overall survival, and time to response and 95% CI will be calculated.
- Major molecular response rate will be defined as the proportion of patients who meet the criteria for MMR at least once after the initiation of study treatment. The analysis will be performed using a 2-sided exact 95% CI for the MMR rate.

### 4.2.4.4 Data Handling Rules for Secondary Endpoint Analyses

In addition to the data handling rules specified in Section 4.2.3.2, the following key data handling rules for the secondary efficacy analyses will be implemented (note that the definition of progression is specified in Attachment A of the protocol).

- Loss of MCyR is defined as meeting any of the following criteria:
  - o Patients entering the trial in PCyR: 2 consecutive cytogenetic assessments ≥ 28 days apart with Ph+ > 0% after achieving a CCyR. Patients with a single cytogenetic assessment with Ph+ > 0% followed by no additional cytogenetic assessments will be also considered as meeting the criteria for loss of MCyR.
  - O Patients entering the trial not in PCyR: 2 consecutive cytogenetic assessments 28 days apart with Ph+ > 35% after achieving a PCyR. Patients with a single cytogenetic assessment with Ph+ > 35% followed by no additional cytogenetic assessments will be also considered as meeting the criteria for loss of MCyR.
- Loss of MaHR (Cohorts C through F) is defined as 2 consecutive hematologic assessments ≥ 28 days apart at which at the criteria for MaHR are not met. Patients with a single hematologic assessment at which the criteria for MaHR are not met followed by no additional hematologic assessments will be also considered as meeting the criteria for loss of MaHR.
- Patients who progress after a single missed or incomplete visit will be considered as having progressed at the visit at which progression was documented.
- Patients who progress after 2 or more missed or incomplete visits will be censored at the last visit at which the response criteria are met. For Cohorts A and B, 2 missed visits will be

defined as more than 182 days between consecutive visits; for Cohorts C-F, 2 missed visits

and a supple of the state of th

## 4.3 Summaries of Data Handling Rules for Primary and Secondary Efficacy Analyses

### Table 6: Summary of Data Handling Rules for Major Cytogenetic Response (MCyR)

Note: all assessments must be after the initiation of study treatment unless otherwise specified.

| | PRIMARY ANALYSIS | SENSITIVITY ANALYSIS 1 | SENSITIVITY ANALYSIS 2 |
|---|---|---|---|
| Population | Per Protocol (Cytogenetic) Population | Treated Population (includes patients with < 20 metaphases examined for baseline cytogenetic assessment) | Treated Population (includes patients with < 20 metaphases examined for baseline cytogenetic assessment) |
| | | cytogenetic assessment) | Patients for whom a <b>positive</b> baseline T315I direct sequencing result is received after the first cytogenetic response assessment (CML patients in CP) or BM assessment (CML patients in AP or BP and Ph+ ALL patients) will be analyzed as T315I |
| | | cial use only | Patients for whom a <b>negative</b> baseline T315I direct sequencing result is received after first cytogenetic response assessment (CML patients in CP) or BM assessment (CML patients in AP or BP and Ph+ ALL patients) will be analyzed as <b>T315I+</b> . |
| MCyR | For patients not in PCyR at study entry (>35% Ph+ cells): 1 assessment of: • 0-35% Ph+ cells with at least 20 | For patients not in PCyR at study entry (>35% Ph+ cells): 1 assessment of: O-35% Ph+ cells with at least 20 | For patients not in PCyR at study entry (>35% Ph+ cells): 1 assessment of: • 0-35% Ph+ cells with at least 20 |
| | metaphases examined | metaphases examined | metaphases examined |
| | OR | OR | OR |
| | • See Table 5 | • See Table 5 | • See Table 5 |
| | For patients in PCyR at study entry (>0% and ≤35% Ph+ cells): 1 assessment of 0% | For patients in PCyR at study entry (>0% and ≤35% Ph+ cells): 1 assessment of 0% | For patients in PCyR at study entry (>0% and ≤35% Ph+ cells): 1 assessment of 0% |
| | Ph+ cells with at least 20 metaphases examined | Ph+ cells with at least 20 metaphases examined | Ph+ cells with at least 20 metaphases examined |
| | -0, | Any time after initiation of study treatment | Any time after initiation of study treatment |
| | ≤ 12 months after initiation of study treatment | | |

| | PRIMARY ANALYSIS | SENSITIVITY ANALYSIS 1 | SENSITIVITY ANALYSIS 2 |
|---|---|---|---|
| Confirmed | For patients not in PCyR at study entry | For patients not in PCyR at study entry | For patients not in PCyR at study entry |
| MCyR | (>35% Ph+ cells): 2 consecutive | (>35% Ph+ cells): 2 consecutive assessments | (>35% Ph+ cells): 2 consecutive assessments |
| | assessments at least 4 weeks apart of: | at least 4 weeks apart of: | at least 4 weeks apart of: |
| | • 0-35% Ph+ cells with at least 20 | • 0-35% Ph+ cells with at least 20 | 0-35% Ph+ cells with at least 20 |
| | metaphases examined | metaphases examined | metaphases examined |
| | OR | OR | OR |
| | • See Table 5 | • See Table 5 | See Table 5 |
| | For patients in PCyR at study entry: 2 consecutive assessments at least 4 weeks apart of 0% Ph+ cells with at least 20 metaphases examined | For patients in PCyR at study entry: 2 consecutive assessments at least 4 weeks apart of 0% Ph+ cells with at least 20 metaphases examined | For patients in PCyR at study entry: 2 consecutive assessments at least 4 weeks apart of 0% Ph+ cells with at least 20 metaphases examined |
| | $\leq$ 12 months after initiation of study | Any time after initiation of study treatment | Any time after initiation of study treatment |
| | treatment | | |

Table 7: Summary of Data Handling Rules for Major Hematologic Response (MaHR)

| | , | | |
|---|---|---|---|
| | PRIMARY ANALYSIS | SENSITIVITY ANALYSIS 1 | SENSITIVITY ANALYSIS 2 |
| Population | Per Protocol (Hematologic) Population | Treated Population (includes patients with baseline bone marrow assessments for which percent blast cannot be determined) | Treated Population (includes patients with baseline bone marrow assessments for which percent blast cannot be determined) Patients for whom a positive baseline |
| | | orly and subject to the | T315I direct sequencing result is received after the first cytogenetic response assessment (CML patients in CP) or BM assessment (CML patients in AP or BP and Ph+ ALL patients) will be analyzed as T315I |
| | | conty and st | patients) will be analyzed as 13151+. |
| MaHR<br>(CHR) | 1 assessment at which all of the following criteria are met: • WBC ≤ ULN • ANC ≥ 1000/mm³ • Platelets ≥ 100,000/mm³ • No blasts or promyelocytes in peripheral blood • BM blasts ≤ 5% • < 5% myelocytes plus metamyelocytes in peripheral blood • Basophils in peripheral blood < 5% • No extramedullary involvement (including no hepatomegaly) | 1 assessment at which all of the following criteria are met: • WBC ≤ ULN • ANC ≥ 1000/mm³ • Platelets ≥ 100,000/mm³ • No blasts or promyelocytes in peripheral blood • BM blasts ≤ 5% • < 5% myelocytes plus metamyelocytes in peripheral blood • Basophils in peripheral blood < 5% • No extramedullary involvement (including no hepatomegaly or splenomegaly) | 1 assessment at which all of the following criteria are met: • WBC ≤ ULN • ANC ≥ 1000/mm³ • Platelets ≥ 100,000/mm³ • No blasts or promyelocytes in peripheral blood • BM blasts ≤ 5% • < 5% myelocytes plus metamyelocytes in peripheral blood • Basophils in peripheral blood < 5% • No extramedullary involvement (including no hepatomegaly or splenomegaly) |
| | $\leq$ 6 months after initiation of study treatment | Any time after initiation of study treatment | ≤ 6 months after initiation of study treatment |

| 1 additional assessment at which all of the following criteria are met, at least 28 days after the first assessment of response: • WBC ≤ ULN • ANC ≥ 1000/mm³ • Platelets ≥ 100,000/mm³ • No blasts or promyelocytes in peripheral blood 1 additional assessment at which all of the following criteria are met, at least 28 days after the first assessment of response: • WBC ≤ ULN • ANC ≥ 1000/mm³ • Platelets ≥ 100,000/mm³ • No blasts or promyelocytes in peripheral blood 1 additional assessment at which all of the following criteria are met, at least 28 days after the first assessment of response: • WBC ≤ ULN • ANC ≥ 1000/mm³ • Platelets ≥ 100,000/mm³ • No blasts or promyelocytes in No blasts or promyelocytes in | |
|---|---|
| <ul> <li>ANC ≥ 1000/mm³</li> <li>Platelets ≥ 100,000/mm³</li> <li>No blasts or promyelocytes in peripheral blood</li> <li>MBC ≤ ULN</li> <li>ANC ≥ 1000/mm³</li> <li>Platelets ≥ 100,000/mm³</li> <li>Platelets ≥ 100,000/mm³</li> <li>No blasts or promyelocytes in</li> <li>No blasts or promyelocytes in</li> </ul> | |
| <ul> <li>&lt; 5% myelocytes plus metamyelocytes in peripheral blood</li> <li>Basophils in peripheral blood &lt; 5%*</li> <li>= 5% myelocytes plus metamyelocytes in peripheral blood</li> <li>= 5% myelocytes plus metamyelocytes in peripheral blood</li> <li>= 5% myelocytes plus metamyelocytes in peripheral blood</li> <li>= Basophils in peripheral blood</li> <li>= Basophils in peripheral blood</li> <li>= Basophils in peripheral blood</li> </ul> | blood<br>< 5%* |
| MaHR (NEL) 1 assessment at which all of the following criteria are met: 1 assessment at which all of the following criteria are met: 1 assessment at which all of the following criteria are met: | ing |
| <ul> <li>WBC ≤ ULN</li> <li>No blasts or promyelocytes in peripheral blood</li> <li>BM blasts ≤ 5%</li> <li>&lt; 5% myelocytes plus metamyelocytes in peripheral blood</li> <li>Basophils in peripheral blood </li> <li>Basophils in peripheral blood </li> <li>No extramedullary involvement (including no hepatomegaly)</li> <li>At least 1 of the following: (i) 20,000/mm³ ≤ platelets &lt; 100,000/mm³; (ii) 500/mm³ ≤ ANC &lt; 10000/mm³</li> <li>WBC ≤ ULN</li> <li>No blasts or promyelocytes in peripheral blood</li> <li>BM blasts ≤ 5%</li> <li>&lt; 5% myelocytes plus metamyelocytes in peripheral blood</li> <li>Basophils in peripheral blood</li> <li>No extramedullary involvement (including no hepatomegaly or splenomegaly)</li> <li>At least 1 of the following: (i) 20,000/mm³ ≤ platelets &lt; 100,000/mm³; (ii) 500/mm³ ≤ ANC &lt; 10000/mm³</li> <li>&lt; WBC ≤ ULN</li> <li>No blasts or promyelocytes in peripheral blood</li> <li>BM blasts ≤ 5%</li> <li>&lt; 5% myelocytes plus metamyelocytes in peripheral blood</li> <li>No extramedullary involvement (including no hepatomegaly or splenomegaly)</li> <li>At least 1 of the following: (i) 20,000/mm³ ≤ platelets &lt; 100,000/mm³ ≤ platelets &lt; 100,000/mm³; (ii) 500/mm³ ≤ 10000/mm³</li> </ul> | blood<br>< 5%<br>ent<br>or<br>ANC |
| ≤ 6 months after initiation of study treatment 1 additional assessment at which all of the following criteria are met, at least 28 days after the first assessment of response: Any time after initiation of study treatment 1 additional assessment at which all of the following criteria are met, at least 28 days after the first assessment of response: ≤ 6 months after initiation of study treatment 1 additional assessment at which all of the following criteria are met, at least 28 days after the first assessment of response: the first assessment of response: | the |

| PRIMARY ANALYSIS | SENSITIVITY ANALYSIS 1 | SENSITIVITY ANALYSIS 2 |
|---|---|---|
| • WBC ≤ ULN | • WBC ≤ ULN | • WBC ≤ ULN |
| <ul> <li>No blasts or promyelocytes in<br/>peripheral blood</li> </ul> | <ul> <li>No blasts or promyelocytes in<br/>peripheral blood</li> </ul> | <ul> <li>No blasts or promyelocytes in<br/>peripheral blood</li> </ul> |
| <ul> <li>&lt; 5% myelocytes plus<br/>metamyelocytes in peripheral blood</li> </ul> | • < 5% myelocytes plus<br>metamyelocytes in peripheral blood | < 5% myelocytes plus<br>metamyelocytes in peripheral blood |
| <ul> <li>Basophils in peripheral blood &lt; 5%</li> </ul> | • Basophils in peripheral blood < 5% | <ul> <li>Basophils in peripheral blood &lt; 5%</li> </ul> |
| • At least 1 of the following: (i) $20,000/\text{mm}^3 \le \text{platelets} < 2$ | • At least 1 of the following: (i) $20,000/\text{mm}^3 \le \text{platelets} < 20,000/\text{mm}^3 \le platel$ | • At least 1 of the following: (i) 20,000/mm <sup>3</sup> \( \le \) platelets < |
| 100,000/mm <sup>3</sup> ; (ii) 500/mm <sup>3</sup> ≤ ANC <1000/mm <sup>3</sup> | 100,000/mm <sup>3</sup> ; (ii) 500/mm <sup>3</sup> \(\leq \text{ANC}\) \(<1000/\text{mm}^3\) | 100,000/mm <sup>3</sup> ; (ii) 500/mm <sup>3</sup> ≤ ANC <1000/mm <sup>3</sup> |

<sup>\*</sup>Refer to protocol amendment 1; basophils in peripheral blood changed from <20% to <5%.

Table 8: Summary of Data Handling Rules for Analysis of Duration of Response†

| CONDITION | ANALYSIS 1 | ANALYSIS 2 | ANALYSIS 3 | ANALYSIS 4 |
|---|---|---|---|---|
| | | | dicar | (Duration of Confirmed<br>Response) |
| No progression or loss of response | Censored at last date patient met criteria for response | Censored at date of last dose of study drug | Censored at date of last dose of study drug | Censored at last date patient met criteria for response |
| Progression or loss of response* any time after a single (unconfirmed) assessment of response | Progression (Duration = Date of relapse – Date of first response assessment) | Progression (Duration = Date of relapse – Date of first response assessment) | Progression (Duration = Date of relapse - Date of first response assessment) | Excluded |
| Progression or loss of response<br>any time after two consecutive<br>assessments of response at least 4<br>weeks apart (confirmation of<br>response) | Progression (Duration = Date of relapse – Date of first response assessment) | Progression (Duration = Date of relapse – Date of first response assessment) | Progression (Duration = Date of relapse – Date of first response assessment) | Progression (Duration = Date of relapse – Date of second response assessment) |
| Progression or loss of response after one missed or incomplete assessment | Progression (Duration = Date of relapse – Date of first response assessment) | Progression (Duration = Date of relapse – Date of first response assessment) | Progression (Duration = Date of relapse – Date of first response assessment) | Censored at last date patient met criteria for response |
| Progression or loss of response<br>after two or more missed or<br>incomplete assessments | Censored at last date patient met criteria for response | Censored at date of last dose of study drug | Progression (Duration = Date of relapse – Date of first response assessment) | Censored at last date patient met criteria for response |
| Initiation of prohibited anti-<br>leukemia therapy (including stem<br>cell transplant) prior to loss of<br>unconfirmed response | Censored at date of initiation of new therapy | Censored at date of initiation of new therapy | Censored at date of initiation of new therapy | Excluded |
| Initiation of prohibited anti-<br>leukemia therapy (including stem<br>cell transplant) prior to loss of<br>confirmed response | Censored at date of initiation of new therapy | Censored at date of initiation of new therapy | Censored at date of initiation of new therapy | Censored at last date patient met criteria for response |

| CONDITION | ANALYSIS 1 | ANALYSIS 2 | ANALYSIS 3 | ANALYSIS 4 (Duration of Confirmed Response) |
|---|---|---|---|---|
| Cohorts A and B: Failure to respond by 12 months after the initiation of study treatment Cohorts C, D, E, and F: Failure to respond by 6 months after the initiation of study treatment | Excluded | Excluded | Included if patient meets criteria for response | Excluded |

<sup>&</sup>lt;sup>†</sup> An additional analysis will be performed defining the duration as the time from the first assessment at which the criteria for response are met until the last assessment at which the criteria for response are met.

Table 9: Summary of Data Handling Rules for Analysis of Major Molecular Response (MMR)

| CONDITION | ANALYSIS 1 | ANALYSIS 2 | ANALYSIS 3 |
|---|---|---|---|
| No baseline result obtained | Non-success | Excluded | Analyze as observed |
| MMR at baseline | Non-success | Excluded | Analyze as observed |
| Detectable levels of BCR-ABL and ABL at baseline followed by Not Detectable levels of BCR-ABL post-baseline | Success | Success | Success |
| Measurement of BCR-ABL or ABL considered to be aberrant upon medical review | Data point will be used for determination of MMR | Data point will be excluded for determination of MMR | Data point will be excluded for determination of MMR |

#### 4.3.1 Subgroup Analyses of the Primary Endpoints and Key Secondary Endpoints

For the primary endpoint and selected key secondary endpoints, subgroup analyses will be performed by key baseline potential prognostic factors. Subgroups will include:

- Age
- Gender
- Race
- Eastern Cooperative Oncology Group (ECOG) performance status
- Geographic Region (US vs. Rest of World [ROW])
- Time Since Diagnosis
- **Mutation Status** 
  - Via Direct Sequencing method
  - Via allele-specific oligonucleotide (ASO) method

    T315I+ vs. T315IT315I status by history
    T315+ vs. T315I
    FKI Exposure
  - o T315I status by history
- Prior TKI Exposure
- Deep performance status orld [ROW])

  Let Sequencing method
  T315I mutation
  Kinase Domain (KD) mutations other than T315I
  No detectable KD mutations
  le-specific oligonucleotide (ASO) method
  T315I+ vs. T315Iatus by history
  315+ vs. T315Iire
  prior TKT
  ) o 2<sup>nd</sup> line (1 prior TKI) vs. 3<sup>rd</sup> line (any 2 prior TKIs) vs. >3<sup>rd</sup> line (any 3 or more prior TKIs)
  - Nilotinib Exposure (Yes/No)
  - Dasatinib Exposure (Yes/No)
  - o Intolerant vs. Resistant (to Dasatinib or Nilotinib)
- BCR-ABL/ABL transcript ratio
- PCvR at baseline
- High-enrolling investigational sites (if applicable)
- Other Disease-Related Prognostic Factors
- T315I and Resistant-Intolerant patients will be pooled within disease groups where applicable (eg, pooling of Cohorts A and B)

#### Treated Patients Not Eligible for Cohorts A-F 4.3.2

Patients who receive study treatment but who are not confirmed to have a detectable baseline T315I mutation by direct sequencing and who are not resistant or intolerant to dasatinib or nilotinib will be analyzed separately according to the data handling rules for primary and secondary efficacy analyses, if applicable.

#### 4.3.3 **Safety Analyses**

All safety analyses will be performed on the safety population, which will include all patients who have received at least one dose of study drug. The safety data from all cohorts will be pooled.

The adverse event incidence rates, as well as the frequency of occurrence of overall toxicity categorized by toxicity grades (severity), will be described. All adverse events starting on or

after the first dose of study treatment will be considered treatment-emergent. In addition, adverse events will be summarized by relatedness to study treatment (in the opinion of the investigator) and action taken with study treatment, including dose modifications, interruptions

Laboratory data results will be standardized and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (NCI CTCAE, v.4.0) criteria when applicable. Change from baseline to the worst on-study result will be summation for these standardized results. Listings of laboratory test results will be summation.

#### 4.3.4 **Study Drug Exposure**

Parameters pertaining to study drug exposure (number of doses, cumulative dose, days from first dose to last dose) will be summarized separately for each cohort. Compliance will also be summarized, including percent compliance, and number of patients with a dose delay or dose reduction.

#### **Exploratory Analyses** 4.3.5

The following exploratory analyses will be performed:



#### 5 REFERENCES

- rems of Use 1. Giles FJ, et al. (2007). Nilotinib therapy after dasatinib failure in patients with imatinibresistant chronic myeloid leukemia (CML) in chronic phase (CP), accelerated phase (AP) or blast crisis (BC). Blood (ASH Annual Meeting Abstracts) 110: Abstract1029.
- 2. Quintas-Cardama A, Kantarjian H, et al. (2007). Dasatinib (BMS-354825) is active in Philadelphia chromosome-positive chronic myelogenous leukemia after imatinib and nilotinib (AMN107) therapy failure. Blood 109(2): 497-499.
- 3. Garg RJ, Kantarjian H, et al. (2009). The use of nilotinib or dasatinib after failure to 2 prior tyrosine kinase inhibitors: long-term follow-up. Blood 114(20): 4361-4368.
- As a phase c ABL mutat, the phase c ABL mutat 4. Muller MC, Cortes J, et al. (2009). Dasatinib treatment of chronic-phase chronic myeloid leukemia: analysis of responses according to preexisting BCR-ABL mutations. Blood